CLINICAL TRIAL: NCT04240080
Title: The Impact of Near-Infrared Vein Mapping on Outcomes and Satisfaction After Botox/Filler Treatment
Brief Title: Impact of Near-Infrared Vein Mapping on Outcomes and Satisfaction After Botox/Filler Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Practice volume was low and resulted in a lack of participant accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William J. Casey, III, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-011561
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Goup (No Intervention): Subjects will undergo clinically indicated facial injection procedures per standard of care without venous mapping
- Intervention Group (Experimental): Subjects will undergo clinically indicated facial injection procedure with pre-procedural facial venous mapping by Accuvein® Veinfinder
  Interventions: Device: Accuvein® Veinfinder

INTERVENTIONS:
Device: Accuvein® Veinfinder — Near-infrared light reflection utilized by healthcare providers to see superficial veins under the skin.
  Arms: Intervention Group

SUMMARY:
Researchers are studying how vein mapping impacts patient outcomes and satisfaction after facial injection procedures.

DETAILED DESCRIPTION:
Facial Botox/filler injections carry risk of puncturing superficial veins, leading to bruising and pain. Our study will investigate the utility of non-invasive vein imaging (specifically near-infrared light reflection) on the incidence of pain/bruising/hematoma and patient satisfaction after facial injections.

The current standard of care for facial injection procedures does not involve any modality of facial venous mapping. Vein mapping is a non-invasive, simple task that takes very little time to conduct. One risk is patient time, however maximum extra time needed will be 5 minutes during the clinical visit. This potential extra time in mind, the benefits far outweigh the risks.

Two cohorts of patients will be prospectively compared following randomization, those who did have pre-procedure venous mapping prior to injection versus those who did not. Data will be analyzed with regard to bruising and swelling following injection, as well as other potential complications such as hematoma or infection, along with patient satisfaction survey information.

ELIGIBILITY:
Inclusion Criteria:

* Patients pursuing aesthetic/therapeutic facial injection procedures (botox/filler)

Exclusion Criteria:

* Patients undergoing aesthetic facial procedures not requiring needle injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | Approximately 7-10 days following the procedure
  Measured using the self-reported FACE-Q satisfaction score, using a scale of 1=definitely disagree and 4=definitely agree

SECONDARY OUTCOMES:
Rate of Bruising/Hematoma | Approximately 7-10 days following the procedure
  Number of subjects to experience bruising/hematoma post facial injection procedure

CONTACTS AND LOCATIONS:
Overall Officials: William Casey III, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials